CLINICAL TRIAL: NCT05566184
Title: The Effect of Modified Pacifier on Pain, Physiological Variables, and Stress Level in Children Connected to Mechanical Ventilators During Vascular Opening
Brief Title: Mechanically Ventilated Children and Pacifiers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Selen Ozakar Akca, Associate Professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HititUS
Record Dates: First submitted 2022-07-12; First posted 2022-10-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Mechanical Ventilation Complication; Pneumonia; Bronchiolitis
Keywords: Mechanical ventilator; Pacifier; Child; Pain; Stress
MeSH Terms: conditions — Pneumonia; Bronchiolitis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified pacifier (Experimental): In the experimental group, a modified pacifier will be given to the child during the procedure and the data will be collected.
  Interventions: Device: Modified pacifier
- Without modified pacifier (No Intervention): Data will be collected without giving the child in the control group a modified pacifier during the procedure.

INTERVENTIONS:
Device: Modified pacifier — In the experimental group, a modified pacifier will be given to the child during the procedure, and the data will be collected. In the application of vascular access to children, a) before the procedure (20 minutes before), b) just before the procedure (20. minutes), c) during the procedure (between 20.-40. minutes), and d) 20 minutes after the procedure (40. minutes). Physiological variables that will be evaluated four times, once for each application, will be observed on the monitor, the FLACC Pain Assessment Scale will be recorded by the researcher and salivary cortisol level will be measured.
  Arms: Modified pacifier

SUMMARY:
Mechanical ventilation is a life support system developed to support or restore normal lung functions. Children who are connected to mechanical ventilator, separation from family in intensive care environment, getting away from the usual home environment, noise of devices, invasive interventions, etc. as a result of many medical diagnosis and treatment procedures, they experience stress because they are exposed to painful stimuli. These painful stimuli are a powerful source of stress and trauma. Stress is a factor that increases the susceptibility to physical and mental tension and illness due to physical, chemical or emotional factors. The stress experienced by children in the Pediatric Care Intensive Unit (PICU) due to painful stimuli can lead to an increase in the secretion of glucocorticoids, especially cortisol, and may cause long-term neurodevelopmental problems and adverse events such as an increase in heart rate, an increase in catabolization and a decrease in oxygen saturation values may occur. Pharmacological and non-pharmacological pain management is required to reduce and minimize pain during short-term, mild to moderately painful procedures in children in the intensive care unit. For this reason, non-nutritive sucking, which is one of the non-pharmacological methods used in infants / children, has vital importance in controlling pain, providing comfort and neurobehavioral control, increasing physiological stability and oxygenation, reducing stress, effective functioning of the digestive system, and reducing the risk of aspiration. Considering the benefits of the pacifier and intubated children between 12-36 months in PICU; Considering the suggestions that they need to calm and soothe themselves, their coordination in sucking and swallowing reflexes is not good, there are risks of aspiration, their weight gain and discharge are prolonged, the physiological stability caused by stress is impaired, and pacifiers can be used up to the age of 3 years, this study was conducted with The aim of this study was to examine the effects of modified pacifier use on pain, physiological variables and stress level in children between the ages of 12-36 months.

DETAILED DESCRIPTION:
Pharmacological and non-pharmacological pain management is required to reduce and minimize pain during short-term, mild to moderately painful procedures in children in the intensive care unit. For this reason, non-nutritive sucking, which is one of the non-pharmacological methods used in infants / children, has vital importance in controlling pain, providing comfort and neurobehavioral control, increasing physiological stability and oxygenation, reducing stress, effective functioning of the digestive system, and reducing the risk of aspiration. The Turkish Neonatology Association (2018) also recommends that sick babies be supported with a pacifier or empty breast feeding method while they are being cared for in the intensive care unit. In the literature many painful procedures (circumcision, vaccination, IV catheterization, lumbar puncture) It is reported that when used during the test, it provides an analgesic effect and reduces stress. This method activates the sucking reflex through a non-opioid mechanism when a pacifier is placed in the child's mouth, creating an endogenous analgesic effect as a result of tactile sensitivity and stimulation of mechanical receptors. Since sucking prevents swallowing, it protects the baby/child against aspiration. At the same time, the use of pacifiers in stressed babies/children with tachycardia provides stability in heart rate and increases oxygenation, allowing the baby to calm down. Behavioral organization such as self-consolation and soothing develops, and the time spent for sleep and alertness levels increase. All these situations provide the baby with less energy consumption, thus causing the baby to be discharged earlier. In the treatment plan of stressed babies/children with poor sucking, swallowing and breathing coordination, it is recommended to use a pacifier as it helps neurobehavioral organization and maturation, and supports calming.

The Baby-Friendly Hospital Initiative, launched by the United Nations International Children's Emergency Fund [UNICEF] in 1990 to promote and support breastfeeding, established the principles of "Ten Steps to Successful Breastfeeding". It was realized that these principles, which rejected the use of pacifiers in the future, did not take into account the separation of the mother and the baby, and it was suggested that this situation should be brought to the agenda. In 2013, the "Ten Steps to Successful Breastfeeding" application was revised and pacifier use was recommended considering the special situations in which the newborn and mother were separated. In the literature and to prevent delays in nutritional development of babies in intensive care units who have to be separated from their mothers. It is strongly recommended to use pacifiers in justified situations to support the development of maturity levels such as motor organization, neuro behavior. However, it is recommended to stop using pacifiers until the age of 3 at the latest. The habit of sucking, which continues after the age of three, can cause displacement of the teeth, deformities in the teeth, gap between the teeth and narrow-high palate structure.

Painful and invasive procedures for follow-up, diagnostic and therapeutic purposes are an inevitable part of care in the intensive care unit. Effective pain and stress management is at the core of nursing care and is based on a comprehensive assessment of the child's pain and stress. Appropriate assessment of pain response and stress level guides treatment. Physiological changes such as increase in heart rate, respiratory rate and intracranial pressure, increase in blood pressure, decrease in oxygen saturation, sweating in the palms of the hands, change in respiratory pattern, differentiation in skin color and pupil size as a result of activation of the sympathetic nervous system following painful stimuli in children. It is also recommended to use the salivary cortisol level in assessing children's stress and to implement the planned intervention in case of stress. Nurses and the interdisciplinary healthcare team have the responsibility to prevent or minimize pain and stress during these procedures. The nurse's being with the patient for a long time can contribute to the healing process by enabling the evaluation and reduction of the patient's pain and stress. Although many studies have been conducted on the assessment of pain and stress in children dependent on mechanical ventilation, there is no study on the use of pacifiers in children dependent on mechanical ventilation. In this study, a pacifier produced from a modified pacifier shield made of polypropylene (PP), a biocompatible polymer with complete ergonomics, adapted to the intubation tube in children connected to mechanical ventilators, will be used. The fact that the pacifier planned to be used in this study is a pacifier evaluated within the scope of the utility model presents the originality of the study. However, it is thought that the use of pacifiers in children who are dependent on mechanical ventilators, who are in a painful and stressful process, will be beneficial in terms of reducing pain and stress in them and thus providing new evidence to nurses about physiological variables.

Considering the benefits of the pacifier and intubated children between 12-36 months in PICU; Considering the suggestions that they need to calm and soothe themselves, their coordination in sucking and swallowing reflexes is not good, there are risks of aspiration, their weight gain and discharge are prolonged, the physiological stability caused by stress is impaired and pacifiers can be used up to the age of 3 years, the hospital where it is planned to work with them is both intensive and neonatal intensive care unit. Since it was observed that sterile gloves were used as pacifiers in the care unit and PICU infants/children to calm them down, this study was planned to be carried out. Although the use of sterile gloves for this purpose seems to be a good method, it is thought that it is not sustainable in terms of continuing the habit of using pacifiers in the future. The aim of this study was to examine the effects of modified pacifier use on pain, physiological variables and stress level in children aged 12-36 months who are dependent on mechanical ventilation.

The research will be conducted in a City Hospital PICU. During the vascular access procedure; 30 children with modified pacifiers will form the study group, and 30 children with no application will form the control group.

In the study, as data collection tools; Introductory Information Form, Ramsay Sedation Scale (RSS), Face, Legs, Activity, Cry, Consolability (FLACC) Pain Assessment Scale, Physiological Variable Follow-up Form, Salivary Cortisol Level Measurement in Stress Assessment tools will be used.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal age is between 12-36 months
* On a mechanical ventilator (intubated and on nasal Continuous Positive Airway Pressure (CPAP) for at least 12 hours)
* According to the RSS, there are 2 and 3 levels of alertness
* The children of the families who agreed to participate in the study

Exclusion Criteria:

* Mechanical ventilator settings change frequently
* Taking neuromuscular blocking drugs
* Receiving high-dose inotropic support (Dopamine and/or Dobutamine 10mcg/kg/hour)
* Pediatric patients receiving medical treatment for chronic pain

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Assesment | 40 minutes
  FLACC (Face, Legs, Activity, Cry, Consolability) Pain Rating Scale: To assess pain in children and adults, Merkel et al. It is an observational behavior scale developed by A.Ş. in 1997. The Turkish validity and reliability of the scale was made. This scale is scored by the researcher through observation.The total score of the scale ranges from 0 to 10. A score of 0 means that the child is calm and pain-free; A score between 1 and 3 indicates that the child has mild pain; A score between 4 and 6 indicates that the child has moderate pain; A score between 7 and 10 represents that the child has a significant discomfort and associated severe pain. The "FLACC Pain Assessment Scale" is the most important data collection method used to determine pain in pediatric patients.

SECONDARY OUTCOMES:
Physiological Variables (Systolic-diastolic blood pressure [mmHg]) | 40 minutes
  Physiological Variable Follow-up Form: One of the parameters to be measured in this form, which was developed by the researcher in line with the literature, is the child's systolic-diastolic blood pressure (mmHg) parameter. In the study, the systolic-diastolic blood pressure (mmHg) of the child will be measured and recorded just before the procedure, during the procedure, and before the vascular access is opened after the procedure.
Physiological Variables (Heart rate [heart beat/min]) | 40 minutes
  Physiological Variable Follow-up Form: One of the parameters to be measured in this form, which was developed by the researcher in line with the literature, is the heart rate (heart beat/min) parameter. In the study, the heart rate (heart beat/min) of the child will be measured and recorded just before the procedure, during the procedure, and before the vascular access is opened after the procedure.
Physiological Variables (Respiration [breaths per/min]) | 40 minutes
  Physiological Variable Follow-up Form: One of the parameters to be measured in this form, which was developed by the researcher in line with the literature, is the respiration (breaths per/min) parameter. In the study, the respiration (breaths per/min) of the child will be measured and recorded just before the procedure, during the procedure, and before the vascular access is opened after the procedure.
Physiological Variables (Oxygen saturation value [%SpO2]) | 40 minutes
  Physiological Variable Follow-up Form: One of the parameters to be measured in this form, which was developed by the researcher in line with the literature, is the oxygen saturation value (%SpO2) parameter. In the study, the oxygen saturation value (%SpO2) of the child will be measured and recorded just before the procedure, during the procedure, and before the vascular access is opened after the procedure.

OTHER OUTCOMES:
Stress Level Assesment | 40 minutes
  Salivary Cortisol Level Measurement in Stress Evaluation: The unit of measurement for salivary cortisol level is Amount of saliva/microliter. Biochemical measurements are used in the evaluation of children's stress behaviors. The most common biochemical measurement used to determine stress hormones, which is one of the physiological changes caused by stress in children, is cortisol. Cortisol level has been found to be a reliable method for assessing pain and stress in children.

REFERENCES:
- [Background] Sonmez-Duzkaya D, The role of the nurse in the prevention of ventilator-associated pneumonia in the pediatric intensive care unit. The Journal of Pediatric Research. 2014; 1(2): 54-61.
- [Background] Beytut D, Başbakkal Z. Sedation evaluation and use of comfort scale in pediatric intensive care. Journal of Intensive Care Nursing. 2013; 17(2): 52-58.
- [Background] Kahraman A, Başbakkal Z. An assessment method for the stress of newborn ınfants: salivary cortisol level. Balıkesir Health Sciences Journal. 2017; 6(3): 136-141.
- [Background] Brummelte S, Grunau RE, Chau V, Poskitt KJ, Brant R, Vinall J, Gover A, Synnes AR, Miller SP. Procedural pain and brain development in premature newborns. Ann Neurol. 2012 Mar;71(3):385-96. doi: 10.1002/ana.22267. Epub 2012 Feb 28. PMID 22374882
- [Background] Valeri BO, Holsti L, Linhares MB. Neonatal pain and developmental outcomes in children born preterm: a systematic review. Clin J Pain. 2015 Apr;31(4):355-62. doi: 10.1097/AJP.0000000000000114. PMID 24866853
- [Background] Cong X, Wu J, Vittner D, Xu W, Hussain N, Galvin S, Fitzsimons M, McGrath JM, Henderson WA. The impact of cumulative pain/stress on neurobehavioral development of preterm infants in the NICU. Early Hum Dev. 2017 May;108:9-16. doi: 10.1016/j.earlhumdev.2017.03.003. Epub 2017 Mar 23. PMID 28343092
- [Background] Coviello C, Popple Martinez M, Drovandi L, Corsini I, Leonardi V, Lunardi C, Antonelli C, Pratesi S, Dani C. Painful procedures can affect post-natal growth and neurodevelopment in preterm infants. Acta Paediatr. 2018 May;107(5):784-790. doi: 10.1111/apa.14222. Epub 2018 Feb 6. PMID 29341252
- [Background] Cignacco E, Hamers JP, Stoffel L, van Lingen RA, Gessler P, McDougall J, Nelle M. The efficacy of non-pharmacological interventions in the management of procedural pain in preterm and term neonates. A systematic literature review. Eur J Pain. 2007 Feb;11(2):139-52. doi: 10.1016/j.ejpain.2006.02.010. Epub 2006 Apr 3. PMID 16580851
- [Background] Ramos MCM, de Candido LK, Costa T, Leite AC, Manzo BF, Duarte ED, Harrison D, Bueno M. Painful procedures and analgesia in hospitalized newborns: A prospective longitudinal study. Journal of Neonatal Nursing. 2019; 25(1): 26-31.
- [Background] Krishnan L. Pain relief in neonates. J Neonatal Surg. 2013 Apr 1;2(2):19. eCollection 2013 Apr-Jun. No abstract available. PMID 26023439
- [Background] Nyqvist KH, Haggkvist AP, Hansen MN, Kylberg E, Frandsen AL, Maastrup R, Ezeonodo A, Hannula L, Haiek LN; Baby-Friendly Hospital Initiative Expert Group. Expansion of the baby-friendly hospital initiative ten steps to successful breastfeeding into neonatal intensive care: expert group recommendations. J Hum Lact. 2013 Aug;29(3):300-9. doi: 10.1177/0890334413489775. Epub 2013 May 31. PMID 23727630
- [Background] Foster JP, Psaila K, Patterson T. Non-nutritive sucking for increasing physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2016 Oct 4;10(10):CD001071. doi: 10.1002/14651858.CD001071.pub3. PMID 27699765
- [Background] Lubbe W, Ten Ham-Baloyi W. When is the use of pacifiers justifiable in the baby-friendly hospital initiative context? A clinician's guide. BMC Pregnancy Childbirth. 2017 Apr 27;17(1):130. doi: 10.1186/s12884-017-1306-8. PMID 28449646
- [Background] Harding CM, Law J, Pring T. The use of non-nutritive sucking to promote functional sucking skills in premature infants: an exploratory trial. Infant. 2006; 2(6): 238-240.
- [Background] Pinelli J, Symington A. Non-nutritive sucking for promoting physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD001071. doi: 10.1002/14651858.CD001071.pub2. PMID 16235279
- [Background] Gederi A, Coomaraswamy K, Turner PJ. Pacifiers: a review of risks vs benefits. Dent Update. 2013 Mar;40(2):92-4, 97-8, 101. doi: 10.12968/denu.2013.40.2.92. PMID 23600033
- [Background] Vu-Ngoc H, Uyen NCM, Thinh OP, Don LD, Danh NVT, Truc NTT, Vi VT, Vuong NL, Huy NT, Duong PDT. Analgesic effect of non-nutritive sucking in term neonates: A randomized controlled trial. Pediatr Neonatol. 2020 Feb;61(1):106-113. doi: 10.1016/j.pedneo.2019.07.003. Epub 2019 Aug 8. PMID 31474462
- [Background] Wu HP, Yang L, Lan HY, Peng HF, Chang YC, Jeng MJ, Liaw JJ. Effects of Combined Use of Mother's Breast Milk, Heartbeat Sounds, and Non-Nutritive Sucking on Preterm Infants' Behavioral Stress During Venipuncture: A Randomized Controlled Trial. J Nurs Scholarsh. 2020 Sep;52(5):467-475. doi: 10.1111/jnu.12571. Epub 2020 Jun 20. PMID 32564489
- [Background] Jenik AG, Vain N. The pacifier debate. Early Hum Dev. 2009 Oct;85(10 Suppl):S89-91. doi: 10.1016/j.earlhumdev.2009.08.025. Epub 2009 Sep 17. PMID 19762175
- [Background] Neiva FC, Leone CR, Leone C, Siqueira LL, Uema KA, Evangelista D, Delgado S, Rocha A, Buhler KB. Non-nutritive sucking evaluation in preterm newborns and the start of oral feeding: a multicenter study. Clinics (Sao Paulo). 2014 Jun;69(6):393-7. doi: 10.6061/clinics/2014(06)05. PMID 24964303
- [Background] Poyak J. Effects of pacifiers on early oral development. Int J Orthod Milwaukee. 2006 Winter;17(4):13-6. PMID 17256438
- [Background] Rocha CR, Verga KE, Sipsma HL, Larson IA, Phillipi CA, Kair LR. Pacifier Use and Breastfeeding: A Qualitative Study of Postpartum Mothers. Breastfeed Med. 2020 Jan;15(1):24-28. doi: 10.1089/bfm.2019.0174. Epub 2019 Dec 20. PMID 31859530
- [Background] Rheel E, Malfliet A, Van Ryckeghem DML, Pas R, Vervoort T, Ickmans K. The Impact of Parental Presence on Their Children During Painful Medical Procedures: A Systematic Review. Pain Med. 2022 May 4;23(5):912-933. doi: 10.1093/pm/pnab264. PMID 34453832
- [Background] Hellhammer DH, Wust S, Kudielka BM. Salivary cortisol as a biomarker in stress research. Psychoneuroendocrinology. 2009 Feb;34(2):163-171. doi: 10.1016/j.psyneuen.2008.10.026. Epub 2008 Dec 18. PMID 19095358
- [Background] Keil MF. Salivary cortisol: a tool for biobehavioral research in children. J Pediatr Nurs. 2012 Jun;27(3):287-9. doi: 10.1016/j.pedn.2012.02.003. Epub 2012 Mar 8. No abstract available. PMID 22405849
- [Background] Condon EM. Psychosocial Influences on Acceptability and Feasibility of Salivary Cortisol Collection From Community Samples of Children. Res Nurs Health. 2016 Dec;39(6):449-462. doi: 10.1002/nur.21744. Epub 2016 Sep 30. PMID 27686043
- [Background] Rolfsjord LB, Bakkeheim E, Berents TL, Alm J, Skjerven HO, Carlsen KH, Mowinckel P, Sjobeck AC, Carlsen KCL. Morning Salivary Cortisol in Young Children: Reference Values and the Effects of Age, Sex, and Acute Bronchiolitis. J Pediatr. 2017 May;184:193-198.e3. doi: 10.1016/j.jpeds.2017.01.064. Epub 2017 Mar 8. PMID 28284475
- [Background] Kara D, Bayrak NA, Volkan B, Ucar C, Cevizci MN, Yildiz S. Anxiety and Salivary Cortisol Levels in Children Undergoing Esophago-Gastro-Duodenoscopy Under Sedation. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):3-6. doi: 10.1097/MPG.0000000000002142. PMID 30169453
- [Background] Dorfman TL, Sumamo Schellenberg E, Rempel GR, Scott SD, Hartling L. An evaluation of instruments for scoring physiological and behavioral cues of pain, non-pain related distress, and adequacy of analgesia and sedation in pediatric mechanically ventilated patients: A systematic review. Int J Nurs Stud. 2014 Apr;51(4):654-76. doi: 10.1016/j.ijnurstu.2013.07.009. Epub 2013 Aug 27. PMID 23987802
- [Background] Curley MA, Wypij D, Watson RS, Grant MJ, Asaro LA, Cheifetz IM, Dodson BL, Franck LS, Gedeit RG, Angus DC, Matthay MA; RESTORE Study Investigators and the Pediatric Acute Lung Injury and Sepsis Investigators Network. Protocolized sedation vs usual care in pediatric patients mechanically ventilated for acute respiratory failure: a randomized clinical trial. JAMA. 2015 Jan 27;313(4):379-89. doi: 10.1001/jama.2014.18399. PMID 25602358
- [Background] Sorce L, Simone S. Pain and Sedation Management in Mechanically Ventilated Children. J Pediatr Intensive Care. 2015 Jun;4(2):64-72. doi: 10.1055/s-0035-1556748. PMID 31110854
- [Background] Ancora G, Lago P, Garetti E, Merazzi D, Savant Levet P, Bellieni CV, Pieragostini L, Pirelli A. Evidence-based clinical guidelines on analgesia and sedation in newborn infants undergoing assisted ventilation and endotracheal intubation. Acta Paediatr. 2019 Feb;108(2):208-217. doi: 10.1111/apa.14606. Epub 2018 Dec 6. PMID 30290021
- [Background] Senayli Y, Ozkan F, Şenaylı A, Bicakci U. Evaluation of postoperative pain in children with FLACC pain scale in Turkish translation. Turkiye Klinikleri Journal of Anesthesiology Reanimation. 2006; 4(1): 1-4.
- [Background] Sılay F, Akyol A. The Turkish adaptation of two measurement tools used in sedation-agitation and pain assessment in intensive care units: a validity and reliability study. Journal of Intensive Care Nursing. 2018; 22(2): 50-65.
- [Background] Crellin D, Harrison D, Santamaria N, Babl FE. Comparison of the Psychometric Properties of the FLACC Scale, the MBPS and the Observer Applied Visual Analogue Scale Used to Assess Procedural Pain. J Pain Res. 2021 Mar 31;14:881-892. doi: 10.2147/JPR.S267839. eCollection 2021. PMID 33833566
- [Background] Verweij LM, Kivits JTS, Weber F. The performance of the heart rate variability-derived Newborn Infant Parasympathetic Evaluation Index as a measure of early postoperative pain and discomfort in infants-A prospective observational study. Paediatr Anaesth. 2021 Jul;31(7):787-793. doi: 10.1111/pan.14188. Epub 2021 May 6. PMID 33811710
- [Background] McCarthy AM, Kleiber C, Hanrahan K, Zimmerman MB, Westhus N, Allen S. Factors explaining children's responses to intravenous needle insertions. Nurs Res. 2010 Nov-Dec;59(6):407-16. doi: 10.1097/NNR.0b013e3181f80ed5. PMID 20962698
- [Background] Redmann AJ, Wang Y, Furstein J, Myer CM 3rd, de Alarcon A. The use of the FLACC pain scale in pediatric patients undergoing adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2017 Jan;92:115-118. doi: 10.1016/j.ijporl.2016.11.016. Epub 2016 Nov 24. PMID 28012511
- [Background] Cabral DM, Antonini SR, Custodio RJ, Martinelli CE Jr, da Silva CA. Measurement of salivary cortisol as a marker of stress in newborns in a neonatal intensive care unit. Horm Res Paediatr. 2013;79(6):373-8. doi: 10.1159/000351942. Epub 2013 Jun 20. PMID 23796826
- [Background] Maas C, Ringwald C, Weber K, Engel C, Poets CF, Binder G, Bassler D. Relationship of salivary and plasma cortisol levels in preterm infants: results of a prospective observational study and systematic review of the literature. Neonatology. 2014;105(4):312-8. doi: 10.1159/000357555. Epub 2014 Mar 5. PMID 24603497